CLINICAL TRIAL: NCT04477629
Title: Belatacept in De Novo Heart Transplantation - Pilot Study
Brief Title: Belatacept in De Novo Heart Transplantation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 22-01135
Record Dates: First submitted 2020-07-16; First posted 2020-07-20 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Heart Transplantation
Keywords: Heart Transplant; Nulojix
MeSH Terms: interventions — Abatacept; Tacrolimus; Mycophenolic Acid; Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: Study population includes first-time Epstein-Barr virus (EBV) seropositive, male and non-pregnant female heart transplant recipients 18 years of age or older, who are able to provide written informed consent for the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Belatacept (Experimental): Participants will receive Belatacept along with an upfront tacrolimus taper Participants will also receive mycophenolate mofetil and corticosteroids are part of standard of care after heart transplant and will follow dosing recommendations as per standard clinical practice.
  Interventions: Drug: Belatacept; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Drug: Corticosteroid

INTERVENTIONS:
Drug: Belatacept — Belatacept will be given in the following way - 10mg/kg IV day 1, 5, end of weeks 2, 4, 8, 12 then 5mg/kg every 4 weeks.
  Other Names: Nulojix
Drug: Tacrolimus — Non-experimental: Tacrolimus will be given in the following way - trough level at month 1, 10-12ng/mL; month 2-3, 6-10ng/mL; month 4-6, 4-6ng/mL; months 7-9 taper off.
  Other Names: Tacrolimus taper
Drug: Mycophenolate Mofetil — Non-experimental: MMF is part of standard of care after heart transplant and will follow dosing recommendations as per standard clinical practice at 500-1500mg twice a day (BID) (dosed to tolerance and effect).
  Other Names: MMF
Drug: Corticosteroid — Non-experimental: CS is part of standard of care after heart transplant and will follow dosing recommendations as per standard clinical practice at a dose no less than 5mg/d.
  Other Names: CS

SUMMARY:
The purpose of this study is to determine if Belatacept is safe to give to adult heart transplant recipients. Belatacept (NULOJIX) is an anti-rejection medication that is available through a prescription from a doctor. In this research study, belatacept is being used in an investigational manner (not for the purpose that it is approved for).

DETAILED DESCRIPTION:
Long-term outcomes after heart transplant remain suboptimal with renal failure and cardiac allograft vasculopathy contributing to morbidity and mortality. Belatacept is Food and Drug Administration (FDA) approved for use in kidney transplant recipients on the basis of two randomized controlled trials, which demonstrated important renal sparing benefits, a reduction in de novo donor-specific antibodies (DSA), and improved long-term outcomes. In this study, ten (10) primary heart transplant recipients will receive belatacept in addition to mycophenolate mofetil, corticosteroids, and a tacrolimus tapering regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female, age ≥18 to ≤75 years
2. Awaiting a primary heart transplant (listed for heart transplant only)
3. Epstein-Barr virus (EBV) IgG seropositive
4. Able to take oral medication and willing to adhere to the belatacept infusion regimen
5. No desensitization therapy prior to transplant
6. Vaccinations should be up to date for hepatitis B, influenza pneumococcal, haemophilus, varicella zoster virus (VZV), measles, mumps and rubella (MMR), and Human Papilloma Virus (HPV) (for participants < 45 years of age) when available
7. Female subjects of childbearing potential must have a negative pregnancy test (serum or urine) prior to randomization
8. Mechanical support or investigational drug trials where the intervention ends at the time of transplantation are permitted
9. Negative virtual crossmatch

Exclusion Criteria:

1. Candidates awaiting multiorgan transplant
2. Estimated glomerular filtration rate (eGFR) < 45 ml/min/m2
3. Candidates with prior organ transplant
4. Candidates actively being treated with immunosuppressive therapies
5. Candidates who have a history of treatment with cytolytic therapy (e.g. anti-thymocyte globulin)
6. Candidates who are intended to be treated with cytolytic therapy in the post-transplant period as induction therapy
7. EBV (IgG) seronegative
8. Active or prior infection with human immunodeficiency virus (HIV), Hepatitis C (HCV), Hepatitis B (HBV)
9. Untreated latent tuberculosis (TB)
10. All potential candidates will be screened prior to enrolment for a history of tuberculosis (chest radiograph and tuberculosis-Interferon Gamma Release Assay (TB-IGRA) or tuberculin skin tests (TST)). Potential candidates with latent TB must be treated prior to study enrolment
11. Prior history of active tuberculosis
12. Prior history of central nervous system infection
13. Known active current viral, fungal, mycobacterial, or other infections excluding driveline infections - potential participants from endemic areas will additionally be screened for histoplasmosis, blastomycosis, coccidioidomycosis, and strongyloidiasis
14. Vaccination with a live vaccine within the past 30 days
15. Malignancy within the last 5 years
16. Any previous treatment with alkylating agents or total lymphoid irradiation
17. Sensitized heart transplant candidates with panel-reactive antibodies (PRA) >50% or those receiving desensitization treatment
18. Prior treatment with belatacept or abatacept
19. History of severe allergic anaphylactic reactions to humanized or murine monoclonal antibodies
20. Treatment with a disease modifying anti-rheumatic drug (DMARD) or other biologic agent (monoclonal antibody) within the past year
21. Treatment with another investigational drug or other intervention at the time of transplant (excluding device or intervention mechanical support or investigational drug trials where the intervention ends at the time of transplant)
22. Potential candidates for whom a calcineurin inhibitor other than tacrolimus (Prograf®) is anticipated after transplant. If during the course of the study, a participant is transitioned to another calcineurin inhibitor due to side effects or inability to achieve stable therapeutic trough levels, they may continue in the study at the discretion of the investigator
23. Any potential participant who remains on mechanical circulatory support for > 72 hours post-transplant will be excluded from the study
24. The need for ongoing high dose vasopressor support > 72 hours post-transplant
25. The need or anticipated need for post-transplant dialysis
26. Platelet count <75,000/mm (within 24 hours prior to transplant)
27. Absolute neutrophil count (ANC) of less than 2000/mm3 within 24 hours prior to transplant
28. Any past or current medical problems or findings on history, physical examination, or laboratory testing, not listed above, that in the opinion of the investigator, may pose additional risk to participation, may interfere with the participant's ability to comply with study requirements, or that may impact the quality or interpretation of study results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-08-06 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of Major Graft-Related Adverse Events | Up to 18 months after transplantation
  Adverse events that will be counted in the total number include: Episodes of acute cellular rejection ≥ 2R/3A, antibody mediated rejection (AMR) ≥ International Society of Heart and Lung Transplantation (ISHLT) AMR 1, hemodynamically compromised rejection, development of cardiac allograft vasculopathy, graft failure occurring ≥ 14 days post-transplant, the need for re-transplant, serious infection requiring inpatient intravenous therapies, post-transplant lymphoproliferative disorder (PTLD), or death.

SECONDARY OUTCOMES:
Change in Estimated Glomerular Filtration Rate (eGFR) | Baseline and 18 months
Percentage of Individuals with Development of De Novo Donor Specific Antibodies (DSA) | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Marlena V. Habal, MD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - NYU Langone Health, New York, New York
  - Columbia University, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided